CLINICAL TRIAL: NCT07152236
Title: A Clinical Study Evaluating the Safety and Efficacy of B7H3 CAR-T Cell Therapy in Patients With B7H3-Positive Solid Tumors
Brief Title: Clinical Study on the Safety and Efficacy of B7H3 CAR T Cells in Patients With B7H3 Positive Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-25-004
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): The administration can be performed via intravenous infusion, either as a single dose or multiple doses, at a dosage ranging from 3×10⁶ to 1×10⁷ CAR-positive T cells per kilogram of body weight, with an allowable deviation of ±20%.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Eligible subjects who successfully passed screening will receive CAR-T cell infusion on Day 0 after lymphodepleting preconditioning chemotherapy.

SUMMARY:
This single-arm, single-center investigator-initiated trial (IIT) evaluates the safety, efficacy, and pharmacodynamic (PD)/pharmacokinetic (PK) profiles of CAR-T cells in patients with advanced solid tumors.

Eligible subjects are followed until 12 months after infusion or until meeting treatment withdrawal criteria, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. The patient fully understands the study procedures and voluntarily signs the informed consent form.
2. Patients diagnosed with tumors that demonstrate positive B7H3 expression in tumor tissues as confirmed by immunohistochemistry (IHC).
3. Presence of at least one extracranial lesion that is measurable according to the RECIST 1.1 criteria;
4. Estimated survival duration of ≥12 weeks;
5. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤1 at baseline;
6. Recovery from prior treatment-related toxicities to a level below Grade 2.
7. Adequate hematopoietic and organ function without severe impairment;
8. Availability of suitable venous access for leukapheresis, with no contraindications to the collection of white blood cells.

Exclusion Criteria:

1. Patients with a history of or currently diagnosed with other malignant tumors;
2. Presence of brain metastases or clinically significant central nervous system (CNS) disorders;
3. Prior treatment within 14 days or five half-lives (whichever is longer) before blood collection for CAR-T preparation that may interfere with lymphocyte expansion;
4. HIV+，HBV，HCV，EBV，CMV.
5. Positive T-cell interferon-gamma release assay or sputum smear for tuberculosis;
6. Documented history or current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonitis, or significant pulmonary dysfunction;
7. History of severe allergic reactions or known hypersensitivity to any component of the investigational drugs used in the study;
8. Severe cardiovascular disease or uncontrolled refractory hypertension, unless deemed stable and non-interfering with the study by the investigator;
9. Severe hepatic or renal dysfunction, or presence of altered mental status;
10. Active autoimmune or inflammatory neurological disorders;
11. Presence of uncontrolled infections requiring systemic antibiotic, antifungal, or antiviral therapy;
12. Receipt of (attenuated) live vaccines within 4 weeks prior to screening;
13. Individuals with a history of alcohol dependence or substance abuse;
14. Pregnant or lactating women.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety | Up to 1 years after CAR-T infusion
  Count the Incidence of adverse events
Effectiveness evaluation | Up to 1 year after CAR-T infusion
  According to the RECIST 1.1 evaluation criteria for the efficacy of solid tumors, the objective response rate (ORR) of all patients after CAR-T treatment, including complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Up to 1 year after CAR-T infusion
  The highest concentration of CAR-T cell expansion in peripheral blood after administration
Pharmacodynamic parameters | Up to 1 year after CAR-T infusion
  The peak values of CAR-T-related cytokines, which include at least IL-6 and IFN-γ.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan Taixin Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No